CLINICAL TRIAL: NCT05451225
Title: Reducing Duration of Untreated Psychosis Through Early Detection in a Large Jail System - Surveys of Correction Officers
Brief Title: Survey of Correction Officers Before and After a Targeted Education Campaign
Acronym: COsurvey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Vera Institute of Justice (Other); University of Illinois at Chicago (Other); University of South Florida (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Compton, Professor of Psychiatry, Columbia University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: NYSPI 7771 - 251050; R34MH117766 (NIH)
Record Dates: First submitted 2022-06-23; First posted 2022-07-11 (Actual); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Work-Related Condition
Keywords: Correction Officers

STUDY DESIGN:
Intervention Model Description: Feasibility and Acceptability Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted Educational Campaign (TEC) for Correction Officers (Experimental): The investigators will implement a Targeted Educational Campaign (TEC) within 3 jails. The TEC is designed to lead to referrals of detainees (previously not detected as having potential mental health concerns) to Correctional Health Services (CHS) by Correction Officers.
  Interventions: Behavioral: Targeted Educational Campaign

INTERVENTIONS:
Behavioral: Targeted Educational Campaign — Correction Officers will be exposed to the Targeted Educational Campaign (TEC) with the aim to increase their knowledge about the early symptoms of psychosis, and how to make a referral to the Correction Health Services staff, their self-efficacy to detect symptoms of psychosis and make referrals, and their expectations about their ability to be successful in making that referral (and for referrals to result in beneficial outcomes).
  Correction Officers will be approached and recruited during roll call and in the staff canteen where they take their meal breaks, or at a time/location agreed upon by the Department of Correction, to complete brief surveys at three different times; pre-exposure, after 6 months, and after 12 months from the beginning of the TEC.

SUMMARY:
The investigators will implement a multifaceted Target Education Campaign (TEC) within the three jails about recognizing early psychotic symptoms and referring to the Correctional Health Services. This campaign will include print materials and targeted trainings for Correction Officers. To develop all aspects of the TEC, the investigators will convene a workgroup, meeting biweekly for the first 6 months, including the entire investigative team, as well as experts at the Center for Practice Innovations (CPI). Depending on the nature of agreed-upon educational materials, the investigators will use specific areas of expertise at CPI for development. Materials will provide specific, actionable, and persuasive messaging about: (1) how to identify select signs of psychosis, (2) how to refer to the Specialized Early Engagement Support Service (SEESS) (in year 2), and (3) the effectiveness of early treatment through coordinated specialty care for early psychosis. Messaging will be continuous in the three jails.

DETAILED DESCRIPTION:
Because Correction Officers in the three jails of interest are critically positioned to influence pathways to care, print materials will be supplemented with professional outreach and education by the SEESS. Roll-call is the approved venue by which all ongoing education happens for Correction Officers. Roll-calls take place at the beginning of each shift (7am, 3pm, 11pm) every day of the week in the same location and last ~ 15 - 20 minutes; all staff starting that shift attend. During roll-call, brief messages (2-3 minutes) will be delivered by the Controlling Captains, which is the standard practice for communicating important information to Correction Officers. Both daytime and overnight shifts will receive the targeted training for the 24 months of the TEC.

The investigators will collect pre-TEC (baseline) and during-TEC (at 6 months and 12 months) data from Correction Officers through brief surveys, which will be used to test changes in mean scores for knowledge, behavioral expectations, and self-efficacy, which are three key constructs from Social Cognitive Theory.

ELIGIBILITY:
Inclusion Criteria:

* Correction Officers;
* over the age of 21

Exclusion Criteria:

* children under the age of 21 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2022-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael T. Compton, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected from this clinical trials research will be deposited into the National Institute of Mental Health Data Archive (NDA). In order to deposit the data, the investigators will use a consent form that allows broad data sharing within the research community. A global unique identifier (GUID) will be created for each research participant using the software that NIMH provides. Dr. Compton and the research coordinator will work with NIMH to create data dictionaries that are relevant to their research. The investigators will share our results, positive and negative, specific to the cohorts and outcome measures studied.
Time Frame: To be determined
Access Criteria: To be determined

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of the study sample took place in 3 jails on Rikers Island in New York City (NYC): Anna M. Kross Center (AMKC), Rose M. Singer Center (RMSC), and the Robert N. Davoren Complex (RNDC).
Pre-assignment Details: Correction officers (COs) were recruited at each of the 3 time points, baseline, 6 months and 12 months, but did not overlap (different COs at each time point) so the recruitment information will not report on a total # enrolled on a continuum (i.e., total number at the beginning, and then how many moved on to 6 months and to 12 months).
Groups:
- Targeted Educational Campaign (TEC) for Correction Officers: The investigators will implement a Targeted Educational Campaign (TEC) within 3 jails at New York City's Rikers Island. The TEC is designed to lead to referrals of detainees (previously not detected as having potential mental health concerns) to Correctional Health Services (CHS) by Correction Officers.
  Targeted Educational Campaign: Correction Officers will be exposed to the Targeted Educational Campaign (TEC) with the aim to increase their knowledge about the early symptoms of psychosis, and how to make a referral to the Correction Health Services staff, their self-efficacy to detect symptoms of psychosis and make referrals, and their expectations about their ability to be successful in making that referral (and for referrals to result in beneficial outcomes).
  Correction Officers will be approached and recruited during roll call and in the staff canteen where they take their meal breaks, or at a time/location agreed upon by the Department of Correction, to complete brief surveys at three different times; pre-exposure, after 6 months, and after 12 months from the beginning of the TEC.
Period: Baseline
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Started | 200
Completed | 200
Not Completed | 0
Period: 6 Months
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Started | 123 (The enrollment reported at 6 months is not sequential to baseline. Different COs were enrolled during this time period.)
Completed | 123
Not Completed | 0
Period: 12 Months
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Started | 128 (The enrollment reported at 12 months is not sequential to baseline and 6 months. Different COs were enrolled during this time period.)
Completed | 128
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Includes all Correction Officers (COs) that were recruited at all time points (baseline, 6 months and 12 months).
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Number analyzed (Participants) | 451
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Correction officers (COs) were recruited at each of the 3 time points, baseline, 6 months and 12 months, but did not overlap (different COs at each time point) so the recruitment information will not report on a total # enrolled on a continuum (i.e., total number at the beginning, and then how many moved on to 6 months and to 12 months).
  years
    COs Recruited at Baseline: number analyzed (Participants) | 200
    COs Recruited at Baseline | 34.2 (8.0)
    COs Recruited at 6 months: number analyzed (Participants) | 123
    COs Recruited at 6 months | 36.1 (6.4)
    COs Recruited at 12 months: number analyzed (Participants) | 128
    COs Recruited at 12 months | 35.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262
  Male | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 185
  Not Hispanic or Latino | 266
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 258
  White | 46
  More than one race | 0
  Unknown or Not Reported | 125
Educational Attainment [Count of Participants; unit: Participants]
  12th grade or less | 19
  Some college | 114
  Completed college | 277
  Graduate training after college | 28
  Unknown | 13
Location of Enrollment [Count of Participants; unit: Participants]
  Jail A | 193
  Jail B | 176
  Jail C | 82

OUTCOME MEASURES:

1. Primary Outcome: Correction Officers' Knowledge at Baseline
Description: Survey-based scores on knowledge/skills at baseline.
  To measure behavioral capability (knowledge/skills), the investigators used the Correction Officers' Behavioral Capability Scale, which has a minimum value of 0 and maximum value of 10. Higher scores mean better knowledge about psychosis and therefore a better outcome.
Time Frame: Baseline
Population: Only 200 Correction Officers (COs) completed this survey at baseline and therefore data exists for only 200 COs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Number analyzed (Participants) | 200
units on a scale | 6.3 (2.5)

2. Primary Outcome: Correction Officers' Knowledge at 6 Months
Description: Survey-based scores on knowledge/skills at 6-months.
  To measure behavioral capability (knowledge/skills), the investigators used the Correction Officers' Behavioral Capability Scale, which has a minimum value of 0 and maximum value of 10. Higher scores mean better knowledge about psychosis and therefore a better outcome.
Time Frame: 6 months
Population: Only 123 Correction Officers (COs) completed this survey at 6 months and therefore data exists for only 123 COs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Number analyzed (Participants) | 123
units on a scale | 7.3 (2.4)

3. Primary Outcome: Correction Officers' Knowledge at 12 Months
Description: Survey-based scores on knowledge/skills at 12-months.
  To measure behavioral capability (knowledge/skills), the investigators used the Correction Officers' Behavioral Capability Scale, which has a minimum value of 0 and maximum value of 10. Higher scores mean better knowledge about psychosis and therefore a better outcome.
Time Frame: 12 months
Population: Only 128 Correction Officers (COs) completed this survey at 12 months and therefore data exists for only 128 COs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Number analyzed (Participants) | 128
units on a scale | 5.3 (2.9)

4. Primary Outcome: Correction Officers' Behavioral Expectations at Baseline
Description: Survey-based scores on behavioral expectations at baseline.
  To measure expectation, the investigators used the Correction Officers' Expectations Scale, which has a minimum value of 8 and a maximum value of 32. Higher scores mean a better outcome.
Time Frame: Baseline
Population: Only 200 Correction Officers (COs) completed this survey at baseline and therefore data exists for only 200 COs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Number analyzed (Participants) | 200
units on a scale | 21.6 (3.1)

5. Primary Outcome: Correction Officers' Behavioral Expectations at 6 Months
Description: Survey-based scores on behavioral expectations at 6-months
  To measure expectation, the investigators used the Correction Officers' Expectations Scale, which has a minimum value of 8 and a maximum value of 32. Higher scores mean a better outcome.
Time Frame: 6 months
Population: Only 123 Correction Officers (COs) completed this survey at 6 months and therefore data exists for only 123 COs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Number analyzed (Participants) | 123
units on a scale | 23.6 (3.7)

6. Primary Outcome: Correction Officers' Behavioral Expectations at 12 Months
Description: Survey-based scores on behavioral expectations at 12 months.
  To measure expectation, the investigators used the Correction Officers' Expectations Scale, which has a minimum value of 8 and a maximum value of 32. Higher scores mean a better outcome.
Time Frame: 12 months
Population: Only 128 Correction Officers (COs) completed this survey at 12 months and therefore data exists for only 128 COs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Number analyzed (Participants) | 128
units on a scale | 21.7 (5.7)

7. Primary Outcome: Correction Officers' Self-Efficacy at Baseline
Description: Survey-based scores on self-efficacy at baseline.
  To measure self-efficacy, the investigators used the Correction Officers' Self-Efficacy Scale, which has a minimum value of 8 and a maximum value of 32. Higher scores mean a better outcome.
Time Frame: Baseline
Population: Only 200 Correction Officers (COs) completed this survey at baseline and therefore data exists for only 200 COs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Number analyzed (Participants) | 200
units on a scale | 26.8 (3.4)

8. Primary Outcome: Correction Officers' Self-Efficacy at 6 Months
Description: Survey-based scores on self-efficacy at 6-months.
  To measure self-efficacy, the investigators used the Correction Officers' Self-Efficacy Scale, which has a minimum value of 8 and a maximum value of 32. Higher scores mean a better outcome.
Time Frame: 6 months
Population: Only 123 Correction Officers (COs) completed this survey at 6 months and therefore data exists for only 123 COs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Number analyzed (Participants) | 123
units on a scale | 27.4 (3.7)

9. Primary Outcome: Correction Officers' Self-Efficacy at 12 Months
Description: Survey-based scores on self-efficacy at 12-months.
  To measure self-efficacy, the investigators used the Correction Officers' Self-Efficacy Scale, which has a minimum value of 8 and a maximum value of 32. Higher scores mean a better outcome.
Time Frame: 12 months
Population: Only 128 Correction Officers (COs) completed this survey at 12 months and therefore data exists for only 128 COs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
Number analyzed (Participants) | 128
units on a scale | 24.5 (5.7)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Targeted Educational Campaign (TEC) for Correction Officers
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT05451225/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT05451225/ICF_002.pdf